CLINICAL TRIAL: NCT07184411
Title: Efficacy of Activities-based Locomotor Training in Children With Cerebral Palsy.
Brief Title: Activities-based Locomotor Training in Children With Cerebral Palsy
Acronym: ENGAGE-CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2245497; 1R15HD119622-01 (NIH)
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy (CP)
Keywords: Cerebral Palsy; Locomotor Training; Physical Therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activities-based locomotor training (AB-LT) (Experimental): Child will participate in a 3-week intensive AB-LT training program. The child will attend the AB-LT session for a total of 3 hours, 5 days a week for 3 weeks. The AB-LT session will consist of 1 hour of walking and standing in a harness on a treadmill, followed by an hour of play-based physical therapy, then followed by a final 1 hour of walking and standing in a harness on a treadmill. All sessions will be run by a licensed physical therapist who is trained in AB-LT.
  Interventions: Other: Activities-based locomotor training
- Usual care (Active Comparator): During this arm, the child will resume or continue their usual therapy schedule, which may include physical therapy, occupational therapy, and/or speech language pathology. No restrictions will be placed on the type or amount of therapy in which the child can participate.
  Interventions: Other: physical therapy

INTERVENTIONS:
Other: Activities-based locomotor training — Activities-based locomotor training involves placing the child in a partial body-weight supported (PBWS) system over a treadmill. The child is given assistance by trained clinicians to attempt standing and walking on the treadmill for 1 hour. The child then participates in play-based activities aimed to foster independence in an overground (regular) environment for 1 hour. The final hour of the 3-hour session is conducted in the PBWS system with a focus on standing and walking.
  Arms: Activities-based locomotor training (AB-LT)
Other: physical therapy — In this intervention, the child will attend their usual physical therapy sessions.
  Arms: Usual care

SUMMARY:
This project aims to improve the quality of life and functional outcomes for young non-ambulatory children with Cerebral Palsy (CP) by investigating the efficacy of an Activities-Based Locomotor Training (AB-LT) program compared to usual care. By targeting the body structures, activities, and participation components of the World Health Organization's International Classification of Functioning, Disability, and Health (ICF) framework, this study seeks to enhance our understanding of neuroplasticity and motor learning in this population, offering a novel approach to rehabilitation. Results from this research will lead to more effective, individualized therapies that improve motor function, reduce disability, and ultimately lower the long-term healthcare needs associated with CP.

ELIGIBILITY:
Inclusion Criteria: To be eligible for this study, the child must be:

* • Able to hold their head upright for 5 seconds when supported at the trunk in sitting (the minimal amount of head control necessary for safe walking on the partial body weight support system during the AB-LT intervention);

  * Non-ambulatory or not walking as primary means of mobility;
  * Willing to attend the AB-LT intervention at Fortis Therapy Center in Dripping Springs, Texas for 3 hours/ day, 5 days/week, for 3 weeks; and
  * Willing to commit to a total of 7 weeks of the study, and to continue their usual care during the time period in which they are not enrolled in the AB-LT intervention.

Exclusion Criteria: The child must not have:

* • Surgery or botulinum toxin injections in the previous 6 months;

  * Uncontrolled epilepsy; and
  * Uncontrolled cardiovascular disease

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Estimated)
Dates: Start 2026-01-11 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure (GMFM-66) | 4 testing sessions: Baseline, end of week 3, end of week 4, end of week 7.
  The GMFM-66 is the gold standard for measuring gross motor function in children with CP. A child's capabilities are scored across five dimensions (66 items), including Lying and Rolling (Dimension A), Sitting (Dimension B), Crawling and Kneeling (Dimension C), Standing (Dimension D), and Walking, Running, and Jumping (Dimension E).

SECONDARY OUTCOMES:
functional near infrared spectroscopy (fNIRS) | 4 testing sessions: Baseline, end of week 3, end of week 4, end of week 7.
  functional near-infrared spectroscopy (fNIRS) is a non-invasive neuroimaging technique that uses infrared light to assess hemodynamic shifts in the prefrontal cortex during movement. It involves wearing a lightweight neoprene headband that contains sensors.
Child Engagement in Daily Life (CEDL) | 4 testing sessions: Baseline, end of week 3, end of week 4, end of week 7.
  The Child Engagement in Daily Life (CEDL) is a survey completed by parents or caregivers of children, 18 months through 12 years of age. The CEDL describes a child's participation in daily activities such as interactions with others, play, and self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ardolino, PhD, PT, Principal Investigator — Baylor University
Locations (1):
- Fortis Therapy Center, Dripping Springs, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified raw data includes child functional near infrared spectroscopy (fNIRS), child functional gross motor ability levels obtained from the Gross Motor Function Measure (GMFM-66), Child Engagement in Daily Life survey data collected from primary caregivers, and parent-reported demographic information.
  Analyzed data that will be shared at the conclusion of the project includes statistical models, and descriptive analysis.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be made available at the time of associated publication or by the end of the project, whichever comes first. Data will be available in REDCap for at least 10 years.